CLINICAL TRIAL: NCT06610617
Title: Neuromodulation of Central Sensory Integration to Improve Postural Control: A Pilot Study in Older Women With Breast Cancer
Brief Title: Neuromodulation of Central Sensory Integration to Improve Postural Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Brendan McNeish, MD, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY24020169
Record Dates: First submitted 2024-09-17; First posted 2024-09-24 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Survivorship; Quality of Life; Cognitive Deficits, Mild
MeSH Terms: conditions — Cognition Disorders; Lymphoma, Follicular | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The interventional study model is a randomized, double-blinded, crossover trial in older taxane treated breast cancer survivors comparing effects of balance between active and sham treatments of a single exposure of transcranial direct current stimulation to the left dorsolateral prefrontal cortex.
  On 4/2/25, after enrollment of the first 4 cancer survivor participants in the randomized trial, the design was modified to allow cancer survivor participants to opt in or out of the tDCS intervention to compare to the cancer free group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Those who receive tDCS on Visit 1 will receive sham stimulation on Visit 2, and those who receive sham on Visit 21and will receive tDCS stimulation on Visit 2. The order of tDCS and sham stimulation is randomized so half of the participants will receive active tDCS first and half will receive tDCS sham. The study member will also be blinded to delivering active or sham tDCS to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active tDCS, then Sham tDCS (Experimental): Stimulation (tDCS) will be delivered in visit 2. Sham will be delivered in visit 3.
  Interventions: Device: transcranial direct current stimulation (tDCS); Device: Sham tDCS
- Sham tDCS, then Active tDCS (Experimental): Sham will be delivered in visit 2. Stimulation (tDCS) will be delivered in visit 3.
  Interventions: Device: transcranial direct current stimulation (tDCS); Device: Sham tDCS
- No Intervention (No Intervention): Participants with a history of cancer and cancer free participants who participated in a single visit without tDCS or sham.

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS designed to facilitate the excitability of the left dlPFC or sham stimulation on separate visits separated by at least one week in random order, using a double-blinded, within-subject crossover design. Electrode placement and current parameters will be optimized to each participant with the goal of generating an average electric field of 0.25 V/m within the left dlPFC. The direct current delivered by any one electrode will not exceed 2.0 mA; the total amount of current from all electrodes will not exceed 4 mA using the Stimweaver algorithm. Each 20-minute session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort
  Arms: Active tDCS, then Sham tDCS; Sham tDCS, then Active tDCS
Device: Sham tDCS — Active sham in which very low-level currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session. This intervention delivers currents and mimics the sensations induced by tDCS, but does not significantly influence cortical tissue.
  Arms: Active tDCS, then Sham tDCS; Sham tDCS, then Active tDCS

SUMMARY:
The objective is to evaluate if neuromodulation of the PFC can acutely improve sensory integration for balance performance in OTTBCS.

DETAILED DESCRIPTION:
Sensory integration required for balance will be measured using the sensory organization test which includes six conditions in which visual and proprioceptive sensory cues are sequentially referenced (i.e. reduced) to stress available sensory information and sensory integration for postural control. Performance on the sensory organization test has been correlated with falls and successful response to balance perturbation. Balance performance will be evaluated by postural sway. Cognitive function will be assessed using the NIH toolbox with a focus on executive function. tDCS will be used to modify PFC excitability and measure its immediate after-effect on balance performance while performing the sensory organization test in OTTBCS. CIPN severity will be evaluated using measurements of distal proprioception. The study sample will be older breast cancer survivors (n=20) diagnosed and treated with taxane chemotherapy after the age of 60 years to avoid heterogeneity due to multiple cancer types, treatments, and sexes.

Outcome measure were removed. Remaining outcome measures were ones that were assessed both before and after tDCS.

ELIGIBILITY:
Inclusion criteria for breast, ovarian and endometrial cancer survivors:

* Women aged 50-85 years
* Breast, ovarian and/or endometrial cancer survivors, stages I-IV
* Completion of taxane chemotherapy treatment. Taxane combined with a history of anthracycline and/or cyclophosphamide is permitted. Active anti-estrogen therapy is permitted. Receiving platin based agents is permitted.
* Ability to walk without an assistive device
* Ability to speak and read English
* Without neurological disease, aside from chemotherapy induced peripheral neuropathy (CIPN) or chemotherapy related cognitive dysfunction (CRCD)
* No history of a other cancer, with the exception that non-melanoma skin cancers are permitted
* Own a device with capability to sync the Fitbit

Inclusion criteria for older cancer-free women:

* Women aged 50-85 years
* Ability to walk without an assistive device
* Ability to speak and read English
* Without neurological disease
* No history of cancer
* Own a device with capability to sync the Fitbit

Inclusion for older, taxane-treated breast, ovarian, and endometrial cancer survivors (OTTBCS) performing a single visit:

* Women aged 50-85 years
* Breast, ovarian and/or endometrial cancer survivors, stages I-IV
* Completion of taxane chemotherapy treatment. Taxane combined with a history of anthracycline and/or cyclophosphamide is permitted. Active anti-estrogen therapy is permitted. Receiving platin based agents is permitted.
* Ability to walk without an assistive device
* Ability to speak and read English
* Without neurological disease, aside from chemotherapy induced peripheral neuropathy (CIPN) or chemotherapy related cognitive dysfunction (CRCD)
* No history of a other cancer, with the exception that non-melanoma skin cancers are permitted
* Own a device with capability to sync the Fitbit

Exclusion criteria for cancer survivors and older women:

* Inability to stand or walk unassisted for 60 seconds
* Hospitalization within the past three months due to acute illness or as the result of a musculoskeletal injury significantly affecting gait or balance
* Any unstable medical condition
* Diagnosis of a gait disorder, Parkinson's disease, Alzheimer's disease or dementia, multiple sclerosis, previous stroke or other neurodegenerative disorder. Cognitive status assessed via the Telephone Interview of Cognitive Status (mTICS). We will exclude those with marked dementia (score<31)
* Chronic vertigo
* Myocardial infarction within the past six months
* Any history of brain or spine surgery, known hearing, visual, or vestibular impairment
* Active chemotherapy, radiation (see below)
* Currently taking anti-epileptic medication
* Known Brain Metastasis

Exclusion for older, taxane-treated breast, ovarian, and endometrial cancer survivors (OTTBCS) performing a single visit:

* Inability to stand or walk unassisted for 60 seconds
* Hospitalization within the past three months due to acute illness or as the result of a musculoskeletal injury significantly affecting gait or balance
* Any unstable medical condition
* Diagnosis of a gait disorder, Parkinson's disease, Alzheimer's disease or dementia, multiple sclerosis, previous stroke or other neurodegenerative disorder. Cognitive status assessed via the Telephone Interview of Cognitive Status (mTICS). We will exclude those with marked dementia (score<31)
* Chronic vertigo
* Myocardial infarction within the past six months
* Known hearing, visual, or vestibular impairment
* Active chemotherapy, radiation (see below)
* Known Brain Metastasis

Additional Criteria for cancer survivors:

* The following criteria is only exclusionary if participant will receive tDCS. Contraindications to transcranial direct simulation (tDCS), including reported seizure within the past 2 years, Currently taking anti-epileptic medication, active use of neuro-active drugs, metal objects anywhere in the head or the neck, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp. Any history of brain or spine surgery
* Active chemotherapy after the first line of 6 cycles is completed will be eligible.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 48 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Equilibrium Score on Sensory Organization Test | 8 months
  The primary outcome measure of Aim 2 will be the change in composite equilibrium score from before and immediately after a single exposure of tDCS or sham stimulation. Briefly, equilibrium score is assessment of postural sway, which can range from 0 to 100, where a lower score indicates more sway and a zero indicates a fall.

SECONDARY OUTCOMES:
Trail Making B test | 2 months
  To evaluate executive function and processing speed. A higher score is better cognitive function.
Digit Symbol Substitution Test | 2 months
  Test to evaluate executive function and processing speed. A higher score is better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan McNeish, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The University of Pittsburgh will promote the development of new research and new investigators by making the data available to outside investigators. The database will include longitudinal demographic, clinical, functional, and physiologic data, from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by University of Pittsburgh.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.

REFERENCES:
- [Background] McNeish BL, Richardson JK, Bell SG, Whitney DG. Chemotherapy-induced peripheral neuropathy increases nontraumatic fracture risk in breast cancer survivors. JBMR Plus. 2021 Jun 10;5(8):e10519. doi: 10.1002/jbm4.10519. eCollection 2021 Aug. PMID 34368609
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Janelsins MC, Heckler CE, Peppone LJ, Kamen C, Mustian KM, Mohile SG, Magnuson A, Kleckner IR, Guido JJ, Young KL, Conlin AK, Weiselberg LR, Mitchell JW, Ambrosone CA, Ahles TA, Morrow GR. Cognitive Complaints in Survivors of Breast Cancer After Chemotherapy Compared With Age-Matched Controls: An Analysis From a Nationwide, Multicenter, Prospective Longitudinal Study. J Clin Oncol. 2017 Feb 10;35(5):506-514. doi: 10.1200/JCO.2016.68.5826. Epub 2016 Dec 28. PMID 28029304
- [Background] Kolb NA, Smith AG, Singleton JR, Beck SL, Stoddard GJ, Brown S, Mooney K. The Association of Chemotherapy-Induced Peripheral Neuropathy Symptoms and the Risk of Falling. JAMA Neurol. 2016 Jul 1;73(7):860-6. doi: 10.1001/jamaneurol.2016.0383. PMID 27183099
- [Background] Winters-Stone KM, Horak F, Jacobs PG, Trubowitz P, Dieckmann NF, Stoyles S, Faithfull S. Falls, Functioning, and Disability Among Women With Persistent Symptoms of Chemotherapy-Induced Peripheral Neuropathy. J Clin Oncol. 2017 Aug 10;35(23):2604-2612. doi: 10.1200/JCO.2016.71.3552. Epub 2017 Jun 6. PMID 28586243
- [Background] Wang AB, Housley SN, Flores AM, Kircher SM, Perreault EJ, Cope TC. A review of movement disorders in chemotherapy-induced neurotoxicity. J Neuroeng Rehabil. 2021 Jan 25;18(1):16. doi: 10.1186/s12984-021-00818-2. PMID 33494755
- [Background] Mirelman A, Herman T, Brozgol M, Dorfman M, Sprecher E, Schweiger A, Giladi N, Hausdorff JM. Executive function and falls in older adults: new findings from a five-year prospective study link fall risk to cognition. PLoS One. 2012;7(6):e40297. doi: 10.1371/journal.pone.0040297. Epub 2012 Jun 29. PMID 22768271
- [Background] Rosano C, Simonsick EM, Harris TB, Kritchevsky SB, Brach J, Visser M, Yaffe K, Newman AB. Association between physical and cognitive function in healthy elderly: the health, aging and body composition study. Neuroepidemiology. 2005;24(1-2):8-14. doi: 10.1159/000081043. PMID 15459503
- [Background] McNeish BL, Dittus K, Mossburg J, Krant N, Steinharter JA, Feb K, Cote H, Hehir MK, Reynolds R, Redfern MS, Rosano C, Richardson JK, Kolb N. Executive function is associated with balance and falls in older cancer survivors treated with chemotherapy: A cross-sectional study. J Geriatr Oncol. 2023 Nov;14(8):101637. doi: 10.1016/j.jgo.2023.101637. Epub 2023 Sep 28. PMID 37776612
- See also: The Effect of Chemotherapy on Balance, Gait, and Falls Among Cancer Survivors: A Scoping Review — https://www.semanticscholar.org/paper/The-Effect-of-Chemotherapy-on-Balance%2C-Gait%2C-and-A-Wechsler-Wood/dbe4e46d46cc2ba3b3049df77273c0a07a455e53